CLINICAL TRIAL: NCT02092961
Title: A Phase IIB, Multi-Centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study of the Efficacy and Safety of Fostamatinib Disodium Monotherapy Compared With Placebo or Adalimumab Monotherapy in Patients With Active Rheumatoid Arthritis: Magnetic Resonance Imaging Sub-Study
Brief Title: Randomised Double-Blind, Placebo-Controlled, Parallel Group Study in Patients With Active Rheumatoid Arthritis:Magnetic Resonance Imaging Sub-Study
Acronym: OSKIRA 4 SS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: AZ decision to discontinue fostamatinib development in RA; rights to fostamatinib returned to Rigel Pharmaceuticals.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4300C00004Sub
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; OSKIRA; fostamatinib; CE-MRI; DCE-MRI
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dosing Group A (Experimental): Oral treatment and subcutaneous injection.
  Interventions: Drug: Fostamatinib; Drug: Placebo of Adalimumab
- Dosing Group D (Active Comparator): Oral treatment and subcutaneous injection.
  Interventions: Drug: Adalimumab; Drug: Placebo of Fostamatinib
- Dosing Group E (Placebo Comparator): Placebo bid for 6 weeks followed by switch to 100 mg fostamatinib bid for 24 weeks, plus placebo subcutaneous injection every 2 weeks.
  Interventions: Drug: Fostamatinib; Drug: Placebo of Fostamatinib; Drug: Placebo of Adalimumab

INTERVENTIONS:
Drug: Fostamatinib — Fostamatinib 100mg twice daily.
  Arms: Dosing Group A; Dosing Group E
Drug: Adalimumab — Adalimumab 40 mg by subcutaneous injection every 2 weeks for 24 weeks.
  Arms: Dosing Group D
Drug: Placebo of Fostamatinib — Placebo bid for 6 weeks.
  Arms: Dosing Group D; Dosing Group E
Drug: Placebo of Adalimumab — Placebo injection once every two weeks.
  Arms: Dosing Group A; Dosing Group E

SUMMARY:
This is a sub-study of the OSKIRA-4 study, (D4300C0004, NCT01264770) to explore alternative and more sensitive modalities for measuring the beneficial effects of syk inhibition with fostamatinib in patients with active RA. This MRI sub-study was reported later than the main study due to recruitment delays at specialist imaging sites and so is registered and presented entirely separately to the main study results.

This study will investigate the impact of treatment on joint activity and damage by assessing synovitis, osteitis, bone erosions and joint space narrowing.

DETAILED DESCRIPTION:
Sub-study to OSKIRA-4: A Phase IIB, Multi-Centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study of the Efficacy and Safety of Fostamatinib Disodium Monotherapy Compared with Placebo or Adalimumab Monotherapy in Patients with Active Rheumatoid Arthritis: Magnetic Resonance Imaging Sub-Study Date: 21 March 2011 Version: 1 Primary objective: Assess the efficacy of fostamatinib in reducing joint synovial disease activity as measured by: - Change from baseline to Week 6 (versus placebo) in OMERACT RAMRIS synovitis score.

ELIGIBILITY:
Inclusion Criteria: -

* Male or female aged 18 and over
* Active rheumatoid arthritis (RA) diagnosed after the age of 16
* Diagnosis within 5 years prior to study visit 1 and inadequate response to treatment with a maximum 2 Disease-Modifying anti-rheumatic drug (DMARD) therapies, or
* diagnosis within 5 years prior to study visit 1 and intolerance to DMARD therapy, or
* diagnosis within 2 years prior to study visit 1 and no previous use of DMARDs
* 4 or more swollen joints and 4 or more tender/painful joints (from 28 joint count)
* Either Erythrocyte Sedimentation Rate (ESR) blood result of 28mm/h or more, or
* C-Reactive Protein (CRP) blood result of 10mg/L or more
* At least 2 of the following:

  * documented history or current presence of positive rheumatoid factor (blood test),
  * radiographic erosion within 12 months prior to study enrolment,
  * presence of serum anti-cyclic citrullinated peptide antibodies (blood test)
  * Presence of at least one swollen hand or wrist joint.
  * Presence of synovitis on baseline MRI scan, defined as at least 1 joint with RAMRIS synovitis score of +1 or greater.

Exclusion Criteria:

* Females who are pregnant or breast feeding
* Poorly controlled hypertension
* Liver disease or significant liver function test abnormalities
* Certain inflammatory conditions (other than rheumatoid arthritis), connective tissue diseases or chronic pain disorders
* Recent or significant cardiovascular disease
* Significant active or recent infection including tuberculosis
* Previously received treatment with a TNF alpha antagonist (including etanercept, certolizumab, adalimumab, infliximab, golimumab) or anakinra or previous treatment with other biological agent including rituximab, abatacept and tocilizumab
* Use of any DMARDs within 6 weeks before first study visit
* Severe renal impairment
* Neutropenia
* Unable to undergo an MRI examination (e.g. presence of a pacemaker, defibrillator, or other implanted metallic device such as anterior interbody cages, aneurysm clip or pedicle screws)
* Known allergy to Gadolinium-based contrast agent,
* Tattoos [in area of examination if contains metallic pigment]
* Likely to require sedation for the procedure
* eGFR less than 55 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2011-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil MacKillop, MD PhD, Study Director — AstraZeneca
Locations (21):
- United States (6):
  - Research Site, Glendale, Arizona
  - Research Site, Paradise Valley, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Brooklyn, New York
  - Research Site, Jackson, Tennessee
  - Research Site, Austin, Texas
- Research Site, Pleven, Bulgaria
- Research Site, Mississauga, Ontario, Canada
- Research Site, Prague, Czechia
- Germany (2):
  - Research Site, Hamburg
  - Research Site, Munich
- Hungary (2):
  - Research Site, Balatonfüred
  - Research Site, Budapest
- Research Site, Amsterdam, Netherlands
- Research Site, Warsaw, Poland
- Research Site, Yaroslavl, Russia
- South Africa (3):
  - Research Site, Durban
  - Research Site, Pretoria
  - Research Site, Stellenbosch
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Oxford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 198 patients were enrolled: 34, 33 and 30 were randomised to Groups A, D and E (33, 28 and 29 received at least 1 dose of IP). Two of the randomised patients were in the main study (D4300C00004).
Pre-assignment Details: A total of 101 patients failed screening.
Groups:
- FOSTA 100 MG PO BID: Dosing Group A
- ADALIMUMAB 40 MG SC: Dosing Group D
- PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID: Dosing Group E
Period: Overall Study
Arm/Group | FOSTA 100 MG PO BID | ADALIMUMAB 40 MG SC | PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID
Started | 33 (Patients who received treatment) | 28 (Patients who received treatment) | 29 (Patients who received treatment)
Randomised But Did Not Receive Treatment | 1 (Study stopped) | 5 (Eligibility criteria not fulfilled/study stopped) | 1 (Eligibility criteria not fulfilled)
Completed | 12 (Number of patients who completed treatment includes patients who had a dose reduction.) | 14 (Number of patients who completed treatment includes patients who had a dose reduction.) | 13 (Number of patients who completed treatment includes patients who had a dose reduction.)
Not Completed | 21 | 14 | 16
Not completed — Not reported | 1 | 0 | 1
Not completed — Study stopped | 13 | 9 | 12
Not completed — Lack of therapeutic response | 2 | 1 | 3
Not completed — Dev. of study specific discont. criteria | 3 | 0 | 0
Not completed — Adverse Event | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOSTA 100 MG PO BID | ADALIMUMAB 40 MG SC | PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID | Total
Number analyzed (Participants) | 33 | 28 | 29 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11.3) | 53 (12.5) | 48 (14.7) | 51 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 21 | 65
  Male | 11 | 6 | 8 | 25
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 24 | 23 | 21 | 68
  Black or African American | 2 | 1 | 4 | 7
  Indian or Pakistani | 5 | 4 | 0 | 9
  Other | 2 | 0 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: OMERACT RAMRIS Synovitis Score - Comparison of Change From Baseline Between Fostamatinib and Placebo or Adalimumab (Van Elteren)
Description: OMERACT RAMRIS synovitis score was based on 8 joints, scored from MRI images, and ranged from 0 to 24 with a smaller value indicating a better clinical condition. Median changes from baseline are shown at each visit (defined as post-baseline minus baseline) with negative values indicative of a better clinical condition. BID = twice daily, CI = confidence interval, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, MRI = magnetic resonance imaging, OMERACT = Outcome Measures in Rheumatoid Arthritis Clinical Trials, PO = orally, RAMRIS = Rheumatoid Arthritis Magnetic Resonance Image Scoring system, SC = subcutaneous.
Time Frame: Baseline, 6 and 24 weeks
Population: The sub-study analysis set includes those patients who received at least 1 dose of investigational product in the MRI sub-study. Patients were analysed by randomised treatment, but only those with available images were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | FOSTA 100 MG PO BID | ADALIMUMAB 40 MG SC | PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID
Number analyzed (Participants) | 33 | 28 | 29
Units on a scale
  6 weeks (n=25, 22, 20) | -1.50 [-3.00 to 0.00] | -0.50 [-1.00 to 0.00] | 0.00 [-0.50 to 1.63]
  24 weeks (n=18, 16, 18) | -0.25 [-3.00 to 1.00] | -1.03 [-2.00 to 0.00] | 0.00 [-2.75 to 1.00]
Statistical Analysis 1: Comparison: FOSTA 100 MG PO BID vs PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID; 6 weeks; Test type: Superiority or Other; p = 0.022, Van Elteren — A negative value for change from baseline in OMERACT RAMRIS synovitis score indicates a better clinical condition; Estimated using the Van Elteren test stratified by DMARD naivety (DMARD naive vs DMARD-IR/intolerant); Treatment difference = -1.75, 90% CI 2-sided [-2.75 to -0.42] — The point estimate for the median difference in change from baseline and associated 90% CI was calculated using the method of unstratified Hodges-Lehmann. A treatment difference <0 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG PO BID vs ADALIMUMAB 40 MG SC; 24 weeks; Test type: Superiority or Other; p = 0.402, Van Elteren — A negative value for change from baseline in OMERACT RAMRIS synovitis score indicates a better clinical condition; Estimated using the Van Elteren test stratified by DMARD naivety (DMARD naive vs DMARD-IR/intolerant); Treatment difference = 0.50, 90% CI 2-sided [-1.00 to 2.00] — [estimate comment as in outcome 1, analysis 1]

2. Other Pre Specified Outcome: OMERACT RAMRIS Osteitis Score - Comparison of Change From Baseline Between Fostamatinib and Placebo or Adalimumab (Van Elteren)
Description: OMERACT RAMRIS osteitis score was based on 25 joints, scored from MRI images, and ranged from 0 to 75 with a smaller value indicating a better clinical condition. Median changes from baseline are shown at each visit (defined as post-baseline minus baseline) with negative values indicative of a better clinical condition. BID = twice daily, CI = confidence interval, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, MRI = magnetic resonance imaging, OMERACT = Outcome Measures in Rheumatoid Arthritis Clinical Trials, PO = orally, RAMRIS = Rheumatoid Arthritis Magnetic Resonance Image Scoring system, SC = subcutaneous.
Time Frame: Baseline, 6 and 24 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | FOSTA 100 MG PO BID | ADALIMUMAB 40 MG SC | PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID
Number analyzed (Participants) | 33 | 28 | 29
Units on a scale
  6 weeks (n=25, 22, 20) | 0.00 [-0.50 to 0.50] | 0.00 [-1.00 to 0.00] | 0.00 [-0.50 to 1.50]
  24 weeks (n=18, 16, 18) | 0.00 [-3.50 to 6.00] | 0.00 [-1.67 to 1.25] | 0.00 [-1.00 to 2.00]
Statistical Analysis 1: Comparison: FOSTA 100 MG PO BID vs PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID; 6 weeks; Test type: Superiority or Other; p = 0.746, Van Elteren — A negative value for change from baseline in OMERACT RAMRIS osteitis score indicates a better clinical condition; Estimated using the Van Elteren test stratified by DMARD naivety (DMARD naive vs DMARD-IR/intolerant); Treatment difference = 0.00, 90% CI 2-sided [-1.00 to 0.50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FOSTA 100 MG PO BID vs ADALIMUMAB 40 MG SC; 24 weeks; Test type: Superiority or Other; p = 0.413, Van Elteren — A negative value for change from baseline in OMERACT RAMRIS synovitis score indicates a better clinical condition; Estimated using the Van Elteren test stratified by DMARD naivety (DMARD naive vs DMARD-IR/intolerant); Treatment difference = 1.00, 90% CI 2-sided [-1.50 to 3.50] — [estimate comment as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Joint Space Narrowing - Comparison of Change From Baseline Between Fostamatinib and Placebo or Adalimumab (Van Elteren)
Description: Joint space narrowing score was based on 20 joints, scored from MRI images and ranged from 0 to 80 with a smaller value indicating a better clinical condition. Median changes from baseline are shown at each visit (defined as post-baseline minus baseline) with negative values indicative of a better clinical condition. BID = twice daily, CI = confidence interval, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, JSN = joint space narrowing, MRI = magnetic resonance imaging, PO = orally, SC = subcutaneous.
Time Frame: Baseline, 6 and 24 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | FOSTA 100 MG PO BID | ADALIMUMAB 40 MG SC | PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID
Number analyzed (Participants) | 33 | 28 | 29
Units on a scale
  6 weeks (n=25, 22, 20) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  24 weeks (n=18, 16, 18) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.00]
Statistical Analysis 1: Comparison: FOSTA 100 MG PO BID vs PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID; 6 weeks; Test type: Superiority or Other; p = 0.491, Van Elteren — A negative value for change from baseline in JSN score indicates a better clinical condition; Estimated using the Van Elteren test stratified by DMARD naivety (DMARD naive vs DMARD-IR/intolerant); Treatment difference = 0.00, 90% CI 2-sided [0.00 to 0.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FOSTA 100 MG PO BID vs ADALIMUMAB 40 MG SC; 24 weeks; Test type: Superiority or Other; p = 0.341, Van Elteren — A negative value for change from baseline in JSN score indicates a better clinical condition; Estimated using the Van Elteren test stratified by DMARD naivety (DMARD naive vs DMARD-IR/intolerant); Treatment difference = 0.00, 90% CI 2-sided [0.00 to 0.00] — [estimate comment as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: OMERACT RAMRIS Erosions Score - Comparison of Change From Baseline Between Fostamatinib and Placebo or Adalimumab (Van Elteren)
Description: OMERACT RAMRIS erosions score was based on 25 joints and ranged from 0 to 250 with a smaller value indicating a better clinical condition. Median changes from baseline are shown at each visit (defined as post-baseline minus baseline) with negative values indicative of a better clinical condition. BID = twice daily, CI = confidence interval, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, MRI = magnetic resonance imaging, OMERACT = Outcome Measures in Rheumatoid Arthritis Clinical Trials, PO = orally, RAMRIS = Rheumatoid Arthritis Magnetic Resonance Image Scoring system, SC = subcutaneous.
Time Frame: Baseline, 6 and 24 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | FOSTA 100 MG PO BID | ADALIMUMAB 40 MG SC | PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID
Number analyzed (Participants) | 33 | 28 | 29
Units on a scale
  6 weeks (n=25, 22, 20) | 0.00 [0.00 to 1.00] | 0.00 [-0.50 to 0.75] | 0.50 [0.00 to 1.00]
  24 weeks (n=18, 16, 18) | 1.00 [0.00 to 3.00] | 0.00 [-0.75 to 0.50] | 1.25 [0.00 to 4.50]
Statistical Analysis 1: Comparison: FOSTA 100 MG PO BID vs PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID; 6 weeks; Test type: Superiority or Other; p = 0.366, Van Elteren — A negative value for change from baseline in OMERACT RAMRIS erosions score indicates a better clinical condition; Estimated using the Van Elteren test stratified by DMARD naivety (DMARD naive vs DMARD-IR/intolerant); Treatment difference = 0.00, 90% CI 2-sided [-0.50 to 0.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FOSTA 100 MG PO BID vs ADALIMUMAB 40 MG SC; 24 weeks; Test type: Superiority or Other; p = 0.053, Van Elteren — A negative value for change from baseline in OMERACT RAMRIS erosions score indicates a better clinical condition; Estimated using the Van Elteren test stratified by DMARD naivety (DMARD naive vs DMARD-IR/intolerant); Treatment difference = 1.25, 90% CI 2-sided [0.50 to 2.50] — [estimate comment as in outcome 1, analysis 1]

5. Other Pre Specified Outcome: DAS-CRP Score - Comparison of Change From Baseline Between Fostamatinib and Placebo or Adalimumab
Description: DAS28-CRP: Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (CRP) and the patient's own assessment. Scores can take any positive value with a lower value indicating a better clinical condition. Mean changes from baseline in DAS28-CRP score are shown at each visit and are presented as decreases from baseline (defined as baseline minus post-baseline) with larger changes indicative of a better clinical condition. ANCOVA = analysis of covariance, BID = twice daily, CRP = C-reactive protein, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, MRI = magnetic resonance imaging, PO = orally, SC = subcutaneous.
Time Frame: Baseline, 6 and 24 weeks
Population: The sub-study analysis set includes those patients who received at least 1 dose of investigational product in the MRI sub-study. Patients were analysed by randomised treatment in accordance with the intention to treat principle.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG PO BID | ADALIMUMAB 40 MG SC | PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID
Number analyzed (Participants) | 33 | 28 | 29
Units on a scale
  6 weeks (n=32, 27, 27) | 1.4 (1.35) [0.00 to 1.00] | 1.1 (1.16) [-0.50 to 0.75] | 0.5 (1.06) [0.00 to 1.50]
  24 weeks (n=20, 19, 17) | 1.1 (1.61) [0.00 to 3.00] | 1.5 (1.44) [-0.75 to 0.50] | 1.6 (1.39) [0.00 to 4.50]
Statistical Analysis 1: Comparison: FOSTA 100 MG PO BID vs PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID; Change from baseline at Week 6. Nonresponder imputation applied following premature withdrawal, or any DMARD initiation, or for 8 weeks following receipt of parenteral steroids, or for patients with no post baseline data. Patients who prematurely withdrew due to project closure have no imputation applied; Test type: Superiority or Other; p = 0.006, ANCOVA; Includes terms for baseline as a continuous covariate and treatment and DMARD naivety (DMARD naive vs DMARD-IR/intolerant) as factors; Least Square Mean Treatment Difference = 0.89, 90% CI 2-sided [0.36 to 1.41]
Statistical Analysis 2: Comparison: FOSTA 100 MG PO BID vs PLACEBO (6 WKS) THEN FOSTA 100 MG PO BID; Change from baseline at Week 24. Nonresponder imputation applied following premature withdrawal, or any DMARD initiation, or for 8 weeks following receipt of parenteral steroids, or for patients with no post baseline data. Patients who prematurely withdrew due to project closure have no imputation applied; Test type: Superiority or Other; p = 0.496, ANCOVA; [statistical method as in outcome 5, analysis 1]; Least Square Mean Treatment Difference = -0.34, 90% CI 2-sided [-1.16 to 0.49]

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: For placebo treated patients time frame includes both placebo(6 weeks) and fostamatinib(18 weeks) treatment. 1 SAE occurred in these treatment arms began during the 6 week placebo treated period
Groups:
- ADALIMUMAB 40 MG: Dosing Group D
- FOSTA 100 MG BID: Dosing Group A
Arm/Group | ADALIMUMAB 40 MG | FOSTA 100 MG BID | PLACEBO (6 WKS) THEN FOSTA 100 MG BID - FOSTA Period | PLACEBO (6 WKS) THEN FOSTA 100 MG BID - Placebo Period
Serious Adverse Events (participants affected / at risk) | 3/28 | 3/33 | 0/22 | 1/29
Other Adverse Events (participants affected / at risk) | 7/28 | 17/33 | 7/22 | 4/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADALIMUMAB 40 MG (N=28) | FOSTA 100 MG BID (N=33) | PLACEBO (6 WKS) THEN FOSTA 100 MG BID - FOSTA Period (N=22) | PLACEBO (6 WKS) THEN FOSTA 100 MG BID - Placebo Period (N=29)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADALIMUMAB 40 MG (N=28) | FOSTA 100 MG BID (N=33) | PLACEBO (6 WKS) THEN FOSTA 100 MG BID - FOSTA Period (N=22) | PLACEBO (6 WKS) THEN FOSTA 100 MG BID - Placebo Period (N=29)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HYPERTENSION (Vascular disorders) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review and comment on results communications prior to publication. Sponsor will be allowed a review period of at least 60 days from submission but can request that publication be delayed for a period up to 6 months. Any reasonable comments made by the sponsor will be incorporated by the PI into the publication.